CLINICAL TRIAL: NCT00431977
Title: DEtection of Subclinical Coronary AtheRosclerosis in diabeTES Using Coronary CT Angiography (DESCARTES Trial)
Brief Title: Validation Study of Coronary CT Angiography as a Screening Tool in Asymptomatic Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: B-0610/038-002
Record Dates: First submitted 2007-02-05; First posted 2007-02-06 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2006-10

CONDITIONS: Coronary Atherosclerosis; Diabetes Mellitus
Keywords: Coronary Atherosclerosis; Diabetes Mellitus
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus

INTERVENTIONS:
Procedure: coronary computed tomography angiography

SUMMARY:
The purpose of this study is to evaluate the prevalence and clinical predictors of subclinical coronary atherosclerosis and to validate the usefulness of coronary CT angiography as a screening tool in asymptomatic patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is the leading cause of death in patients with diabetes. Patients with diabetes are known to have silent myocardial ischemia more frequently than those without diabetes. Furthermore, CAD in patients with diabetes frequently manifested in advance stage, and morbidity and mortality are higher than those without diabetes. Early screening and treatment of CAD in asymptomatic patients with diabetes might reduce high morbidity and mortality.

In recent advance in technology, coronary CT angiography makes it more accurately and easier in detecting CAD not only in symptomatic patients but also in asymptomatic population. In asymptomatic population, coronary CT angiography could detect subclinical coronary atherosclerosis with high sensitivity and specificity. However, there is a paucity of information on the role of coronary CT angiography as a screening method in high risk asymptomatic population, i.e. asymptomatic patients with diabetes.

Therefore in our study, we will evaluate the prevalence and clinical predictors of subclinical coronary atherosclerosis and to validate the usefulness of coronary CT angiography as a screening tool in asymptomatic patients with type 2 diabetes mellitus.

In this study, we will recruit asymptomatic patients with diabetes. At the time of enrollment, patients will be randomly assigned to coronary CT angiography group or control group using web-based randomization table. One-half of patients will be assigned to coronary CT angiography imaging and follow-up, whereas the other half will be randomized to medical treatment and follow-up only.

When the patients are eligible for study, investigators will give information about the study and obtain written consent. The presence of chest pain symptom will be screened with Rose questionnaire. Medical history and physical examination will be performed, and baseline laboratory work-up will be performed. Investigators will evaluate the status of diabetic complication (retinopathy/nephropathy/cardiac autonomic neuropathy).

After initial clinical and laboratory evaluation, all patients will be followed for adverse cardiac events for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Age 50 ~ 75 years

Exclusion Criteria:

* angina pectoris or anginal equivalent symptoms
* insulin pump user or history of ketoacidosis
* history of myocardial infarction, heart failure, or coronary revascularization
* electrocardiographic evidence of Q-wave myocardial infarction, ischemic ST- segment or T-wave changes, or complete left bundle branch block
* uncontrolled arrythmia
* hypersensitivity to contrast dye
* renal failure
* uncontrolled arrythmia
* hypersensitivity to contrast dye
* renal failure

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2006-11; Study Completion 2012-12

PRIMARY OUTCOMES:
Myocardial infarction
Late revascularization therapy
Cardiac death

SECONDARY OUTCOMES:
Early revascularization therapy
Other procedure (i.e. peripheral vascular procedure)
All-caused death

CONTACTS AND LOCATIONS:
Overall Officials: Huk-Jae Chang, MD, PhD, Study Director — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang hospital, Sungnam-si, Gyeonggi-do, South Korea